CLINICAL TRIAL: NCT06303843
Title: The Effect of Electric Ride-On Cars Use During Transport to the Operating Theatre on Preoperative Anxiety in Children Undergoing Elective Ambulatory Surgery: A Randomised Controlled Trial
Brief Title: The Effect of Electric Ride-On Cars Use During Transport to the Operating Theatre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13.04.2023
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Preoperative Anxiety; Pediatric Surgery
MeSH Terms: conditions — Anxiety Disorders | interventions — Parturition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Transfer to the operating theatre with an electric ride-on car
  Interventions: Other: Transfer with an electric ride-on car
- Controlled group (No Intervention): Transfer to the operating theatre with a paediatric trolley

INTERVENTIONS:
Other: Transfer with an electric ride-on car — The children in the experimental group will be transported to the operating theatre by a electric ride-on car.
  Arms: Intervention group

SUMMARY:
The aim of our study was to evaluate the effect of the use of a electric ride-on car during transport to the operating theatre on preoperative anxiety in children undergoing elective ambulatory surgery. As a distraction method, children in the experimental group will be introduced to the operating theatre with a electric ride-on car. Yale Modified Preoperative Anxiety Scale Child Form will be used to evaluate anxiety. The sample size was determined as 118 as a result of power analysis. 59 children will be included in the experimental group and 59 children in the control group.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Being between 2-10 years old,
* Less than 35 kg (according to the manufacturer's instructions for ride-on battery cars),
* To undergo elective surgery,
* Volunteering to participate in the study.

Exclusion Criteria:

* having cognitive or physical disabilities that may prevent riding a electric ride-on car
* premedication before surgery

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Perioperative anxiety | 30 minutes
  Yale Modified Preoperative Anxiety Scale Child Form

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University Training and Research Hospital, Uşak, Turkey (Türkiye)